CLINICAL TRIAL: NCT00997971
Title: Phase 3 Safety Study of a Partially Hydrolyzed Rice Protein Formula in Healthy Infants
Brief Title: Growth, Tolerance in Healthy Infants Fed a Partially Hydrolyzed Rice Protein
Acronym: Rose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sodilac (Industry)
Responsible Party: Pr Jean-Philippe Girardet (Principal investigator), Hôpital d'enfants Armand Trousseau
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ROS-CL3-001
Record Dates: First submitted 2009-09-14; First posted 2009-10-20 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Growth; Allergy
Keywords: Hydrolysed rice protein formula; Cow's milk protein allergy; Infant formula; Gastrointestinal tolerance
MeSH Terms: conditions — Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modilac Rose 1 (Experimental): Infant formula with partially hydrolysed rice protein
  Interventions: Other: Modilac Rose 1

INTERVENTIONS:
Other: Modilac Rose 1 — Infant formula used for non-breastfed children

SUMMARY:
The purpose of this study is to assess growth and global tolerance in healthy new born infants with minor gastrointestinal troubles and/or allergic risk, fed an experimental partially hydrolyzed rice protein infant formula.

DETAILED DESCRIPTION:
This objective will result in the study of non-inferiority of the experimental formula in terms of variation of weight compared with growth curves after 3 to 6 months of exclusive regime with the experimental formula.

Parents provide informed written consent.

4 visits are forecasted in pediatric surgeries: V1(inclusion), V2 (2 months), V3 (4 months) and V4 (6 months). The last visit corresponds to the beginning of the food diversification decided by the pediatrician. Ideally it takes place at 6 months. If the food diversification starts at 4 months, then V3 and V4 constitute the same last visit.

ELIGIBILITY:
Inclusion Criteria:

* Term health infants with gestational age ranging from 37 to 42 weeks
* Infants less than 1 month old
* Non breastfed children at the inclusion
* Growth parameter normal
* Apgar score > 5 to 7 minutes
* Change in the formula because of digestive troubles (colics, gas, regurgitation) or risks of allergy
* Absence of metabolic, nervous or digestive troubles
* Absence of digestive haemorrhage, apnea or dizzy turn

Exclusion Criteria:

* Partial breastfed children
* Infants presenting a cow's milk protein allergy
* Infants currently participating in another trial
* Infants presenting an organic disease involving medicinal or surgical treatment

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Growth parameters | 2nd, 4th and 6th months

SECONDARY OUTCOMES:
Clinical Tolerance | 3 days before the 2nd and 6th months
Atopic diseases (eczema atopic, asthma) | 2nd and 6th months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Girardet, PhD, Principal Investigator — Hôpital d'enfants Armand Trousseau
Locations (9):
- France (9):
  - Aix-les-Bains
  - Asnières
  - Besançon
  - Boulogne-Billancourt
  - Caen
  - Écully
  - Lyon
  - Meaux
  - Saint-Priest-en-Jarez